CLINICAL TRIAL: NCT03780348
Title: A Novel Low-Cost Tool for a More Efficient and Reliable Weight-for-Height/Length Assessment
Acronym: Yared's-tool
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: JSI Research & Training Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: JSI R&T #18-46
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Severe Acute Malnutrition; Wasting
Keywords: Weigh-for-Height/Length; Assessment
MeSH Terms: conditions — Severe Acute Malnutrition; Cachexia

STUDY DESIGN:
Intervention Model Description: Children will be assigned for nutrition status assessment to either of the two groups that use the 'new' or the 'existing' assessment method
Who Masked: Participant, Care Provider, Investigator
Masking Description: The caregivers of the children, the care provider linking the children to either of the groups and the investigator will not know which group each child is joining and which group is using which method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- New Method (Experimental): 'New' weight-for-height method will be used to assess children assigned to this arm
  Interventions: Diagnostic Test: New Method
- Existing Method (Active Comparator): 'Existing' weight-for-height method will be used to assess children assigned to this arm
  Interventions: Diagnostic Test: Existing Method
- Health Extension Workers (Experimental): Health Extension workers will do weight-for-height assessment using the new method
  Interventions: Diagnostic Test: New Method

INTERVENTIONS:
Diagnostic Test: New Method — A 'new' WHZ tool will be used to assess children.
  Arms: Health Extension Workers; New Method
Diagnostic Test: Existing Method — 'Existing' WHZ tools will be used to assess children
  Arms: Existing Method

SUMMARY:
Weight-for-height/length z-score is one of the indicators used to diagnose acute malnutrition. In the existing method, the assessment involves three steps and takes significant time with a wider room for errors. A new tool is developed to address these drawbacks. A preliminary testing done show encouraging results, but a more robust study is needed. This research will b done with the objective of comparing diagnostic efficiency and reliability of the 'new' method against the 'existing' one using a diagnostic randomized clinical trial method.

DETAILED DESCRIPTION:
Acute malnutrition is a major underlying and direct cause of child death. Weight-for-height/length z score (WHZ) is one of the indicators used to assess nutritional status of children. In the existing method, the assessment involves three steps; measuring height, measuring weight and deciding WHZ using a reference graphs or tables. The assessment takes significant time and has wider room for errors. Due to these drawbacks, it is not used at community level where regular active finding takes place.

A new tool is developed to address these drawbacks. It reduces the steps to two aiming at reducing errors and saving time and energy. This study will compare efficiency and reliability of WHZ assessments done with the new tool against the existing method using a diagnostic randomized clinical trial.

Trained health workers will do WHZ assessments in under five children mobilized for nutrition screening program. The 'average time' needed and proportions of 'classification errors' will be compared between the new and the existing methods. Assessments done by two anthropometry experts will be used as gold standard.

The study will determine the gains of the new tool and can potentially change the global practice and help early detection of huge number of wasted children that are being missed.

ELIGIBILITY:
Inclusion Criteria:

* All children under five years of age living in the study area.

Exclusion Criteria:

* Children for whom weigh-for-height assessments can not be done due to physical deformities and disabilities.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 510 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Reliability | In 3 months
  Proportion of 'assessment errors' between the groups will be compared against that of the gold standard (i.e the assessment done by two experts for each child'
Efficiency of assessment | in 3 months
  The average time needed to complete WHZ assessments using the 'new' method will be compared with that of the 'existing' method
Reliability of WHZ assessments done by community Health Extension Workers | in 3 months
  Proportion of 'assessment errors' by health-extension workers will be compared with that of the 'nurses' and the 'experts'

CONTACTS AND LOCATIONS:
Overall Officials: Yared A Fantaye, MD, MPH, Principal Investigator — JSI Training and Research Institute, Inc.

IPD SHARING:
Plan to Share IPD: No
Nutrition assessment data is sensitive for the country and it can only be shared if the regional health bureau allows. It needs time to get their decision

REFERENCES:
- [Background] Grellety E, Golden MH. Severely malnourished children with a low weight-for-height have a higher mortality than those with a low mid-upper-arm-circumference: I. Empirical data demonstrates Simpson's paradox. Nutr J. 2018 Sep 15;17(1):79. doi: 10.1186/s12937-018-0384-4. PMID 30217205
- [Background] Grellety E, Golden MH. Severely malnourished children with a low weight-for-height have a higher mortality than those with a low mid-upper-arm-circumference: III. Effect of case-load on malnutrition related mortality- policy implications. Nutr J. 2018 Sep 15;17(1):81. doi: 10.1186/s12937-018-0382-6. PMID 30217201
- [Background] Laillou A, Prak S, de Groot R, Whitney S, Conkle J, Horton L, Un SO, Dijkhuizen MA, Wieringa FT. Optimal screening of children with acute malnutrition requires a change in current WHO guidelines as MUAC and WHZ identify different patient groups. PLoS One. 2014 Jul 1;9(7):e101159. doi: 10.1371/journal.pone.0101159. eCollection 2014. PMID 24983995
- [Background] Pelletier D, Haider R, Hajeebhoy N, Mangasaryan N, Mwadime R, Sarkar S. The principles and practices of nutrition advocacy: evidence, experience and the way forward for stunting reduction. Matern Child Nutr. 2013 Sep;9 Suppl 2(Suppl 2):83-100. doi: 10.1111/mcn.12081. PMID 24074320